CLINICAL TRIAL: NCT05029375
Title: The Role of Parental Insightfulness in Enhancing the Acquisition of Social Skills in Young Children With ASD, Following a Parent Mediated Intervention
Brief Title: Parental Insightfulness and the Acquisition of Social Skills in Children With ASD.
Acronym: ASD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bar-Ilan University, Israel (Other)
Collaborators: Israel Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 205698
Record Dates: First submitted 2021-08-12; First posted 2021-08-31 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2022-03

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism, Random Clinical Trial, parental insightfulness
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: two parallel intervention groups differing in parental involvement
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- immediate parental involvement (Experimental): Parental involvement in training is parallel to children's training
  Interventions: Behavioral: PEERS® for Preschoolers
- delayed parental involvement (Experimental): Parental involvement in training will be given at the end of the children's training
  Interventions: Behavioral: PEERS® for Preschoolers

INTERVENTIONS:
Behavioral: PEERS® for Preschoolers — P4P is a 16-week manualized social skills treatment program, adapted from an existing empirically supported social skills intervention for young children with autism
  Other Names: P4P

SUMMARY:
Parental Insightfulness (PI), promotes the development of the child's socio-emotional competence and her ability to have productive and sustaining relationships. PI is even more central in the case of young children with ASD, who struggle to socially communicate their needs and their mental and emotional states. PI's effects on the child's peer-interaction have not been tested and Since parents play a central role in intervention programs for their children with ASD, examining modifiable parent factors as mediators and moderators of treatment effectiveness could contribute to this line of research. The proposed study aims to test how pre intervention PI and intervention-related changes in PI affect parents' ability to support their children in the acquisition of peer-interaction skills. Using the PEERS for Preschoolers (P4P) program, the study will examine the effect of PI and parental involvement in a social skills intervention on children's acquisition and maintenance of social skills.

DETAILED DESCRIPTION:
Parental Insightfulness (PI), the ability to see things from the child's point of view and to think about the motives that underlie the child's behavior, promotes the development of the child's socio-emotional competence and her ability to have productive and sustaining relationships. PI may be even more central in the case of young children with Autism Spectrum Disorder (ASD), who struggle to socially communicate their needs and their mental and emotional states. Previous research showed PI predicts adaptive child functioning and demonstrated the merit of PI both as a moderator and as a mediator of treatment outcomes in interventions that aim to promote PI and parent-child interaction. However, PI's effects on the child's peer-interaction have not been tested. Intervention research in ASD has evolved from the examination of treatment effectiveness to the pursuit of treatment mediators and moderators, that could be utilized for treatment individualization. Since parents play a central role in intervention programs for their children with ASD, examining modifiable parent factors as mediators and moderators of treatment effectiveness could contribute to this line of research. The proposed study aims to test how pre intervention PI and intervention-related changes in PI affect parents' ability to support their children in the acquisition of peer-interaction skills. Using the PEERS for Preschoolers (P4P) program, a parent assisted social skills training program for young children with ASD, the study will examine the effect of PI and parental involvement in a social skills intervention on children's acquisition and maintenance of social skills.

These aims will be tested in the following ways: 1) A randomized controlled trial will compare the effects of the parent-mediated P4P program to those of a P4P program with minimal parent involvement (P4P-mpi) on the outcome and the maintenance of gains in child social skills and on PI. 2) an examination of the role of pretreatment PI as a moderator of children's intervention-related social skills gains and their maintenance, and 3) an examination of the role of treatment related change in PI as a mediator of children's intervention-related social skills gains and their maintenance.

The trial will include 80 young children with ASD, aged 4-7, and their parents, who will be randomized into a P4P treatment group and a P4P-mpi control group. Participants will be tested pre- and post- a 16-week intervention period, as well as 10 weeks later, for follow up. Measures will include a behavioral microanalytic assessment of a peer play interaction and parental insightfulness assessment, a parental reflective functioning questionnaire, and social skills questionnaires filled out by parents and teachers. This study may promote the yet limited research on parent-mediated social skills interventions in young children with ASD and shed light on the role of parental insightfulness in children's treatment-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Autism spectrum disorder
* no cooccurring intellectual impairment

Exclusion Criteria:

* severe behavioral problems

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 85 (Estimated)
Dates: Start 2021-08-28 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Behavioral peer interaction measurement | Immediate post intervention assessment
  The interaction will be videotaped and microanalytically coded for frequency and duration of child behaviors, using a designated computerized system
Insightfulness Assessment | Immediate post intervention assessment
  IA (Insightfulness Assessment) transcripts are scored on ten 9-point rating scales The IA (Insightfulness Assessment) provides a classification of the parent's insightfulness as either established (i.e., positively insightful) or emerging (i.e., non-insightful)
Behavioral peer interaction measurement | 10 weeks post intervention (follow up) assessment
  The interaction will be videotaped and microanalytically coded for frequency and duration of child behaviors, using a designated computerized system
Insightfulness Assessment | 10 weeks post intervention (follow up) assessment
  IA (InsightfulneIA (Insightfulness Assessment) transcripts are scored on ten 9-point rating scales ss Assessment) transcripts are scored on ten 9-point rating scales

SECONDARY OUTCOMES:
Social Responsiveness Scale-second edition (Constantino & Gruber, 2012) | Immediate post intervention assessment
  T scores can be computed for each subscale as well as for the total questionnaire, and for a social communication index. Minimun value is 1, maximum value is 4. higher scores mean worse outcome
Social Responsiveness Scale-second edition (Constantino & Gruber, 2012) | 10 weeks post intervention (follow up) assessment
  T scores can be computed for each subscale as well as for the total questionnaire, and for a social communication index. Minimun value is 1, maximum value is 4. higher scores mean worse outcome
The Social Skills Improvement System (SSIS; Gresham & Elliott, 2008) | Immediate post intervention assessment
  Two standard composite scales can be computed for Social Skills and Behavior Problems. Minimun value is 1, maximum value is 4. higher scores mean better outcome
The Social Skills Improvement System (SSIS; Gresham & Elliott, 2008) | 10 weeks post intervention (follow up) assessment
  Two standard composite scales can be computed for Social Skills and Behavior Problems. Minimun value is 1, maximum value is 4. higher scores mean better outcome
Quality of Play Questionnaire (QPQ; Frankel & Mintz, 2011). | Immediate post intervention assessment
  An Engagement Scale measures the extent that the child engaged in talk and physical interaction with the peer, and a Conflict Scale measures the degree of conflict between peers during the last play date. Minimun value is 0, maximum value is 3. higher scores mean better outcome
Quality of Play Questionnaire (QPQ; Frankel & Mintz, 2011). | 10 weeks post intervention (follow up) assessment
  An Engagement Scale measures the extent that the child engaged in talk and physical interaction with the peer, and a Conflict Scale measures the degree of conflict between peers during the last play date. Minimun value is 0, maximum value is 3. higher scores mean better outcome
The Parental Reflective Functioning Questionnaire (PRFQ; Luyten, Mayes, Nijssens & Fonagy, 2017). | Immediate post intervention assessment
  Items are rated on a 7-point Likert scale. Minimun value is 1, maximum value is 7. higher scores mean better outcome
The Parental Reflective Functioning Questionnaire (PRFQ; Luyten, Mayes, Nijssens & Fonagy, 2017). | 10 weeks post intervention (follow up) assessment
  Items are rated on a 7-point Likert scale. Minimun value is 1, maximum value is 7. higher scores mean better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Ofer Golan, Phd, Principal Investigator — Bar Ilan Univercity
Locations (1):
- Bar-Ilan University, Ramat Gan, Israel